CLINICAL TRIAL: NCT05295238
Title: Purpose in Life Renewal for Adults Who Experienced COVID-19 Illness
Brief Title: Compass Course: COVID-19
Acronym: CC-COVID
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allina Health System (Other)
Responsible Party: Principal Investigator, Mary Radomski, Senior Scientific Advisor, Allina Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 1860339
Record Dates: First submitted 2022-03-23; First posted 2022-03-25 (Actual); Last update posted 2024-07-17 (Actual); Status verified 2024-07

CONDITIONS: COVID-19
Keywords: Purpose in Life
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Compass Course (Experimental): Four groups of up to 12 participants (48 total) will receive the study intervention during Spring and Fall 2022. All participants will complete study questionnaires before and after the sessions.
  Interventions: Behavioral: Compass Course

INTERVENTIONS:
Behavioral: Compass Course — An 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention, called the Compass Course is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in their daily lives.

SUMMARY:
A group of clinicians and researchers developed an 8-session group intervention that integrates education, support, self-reflection, and action-expectation to help people reaffirm or reconstruct self-grounded purpose after significant life events/transitions. The 8 sessions extend over 2-3 months, with 7 weekly sessions and the final session 1 month after Session 7. The intervention, called the Compass Course is structured around the 6 dimensions of flourishing (autonomy, self-acceptance, personal growth, relationships, purpose in life, external mastery), the goal of which is to help people enact behaviors that move them forward in reframing a sense of self and reaffirming or reconstructing a sense of purpose in their daily lives. Participating in this research will involve an introduction session, where informed consent will be obtained, followed by the 8-session intervention for 9 sessions in total.

A team composed of researchers from Courage Kenny Rehabilitation Institute (CKRI) propose to recruit a convenience sample of individuals who were hospitalized with COVID-19 to evaluate the efficacy of administering the Compass Course to a novel population, to improve psychological well-being, engagement in everyday activities, and purpose in life.

A focus group will be scheduled 2 months after the completion of the Compass Course. This session is composed of brief questionnaires and designed to obtain post-course data to help evaluate the Compass Course intervention.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 80 years of age;
* Are part of the Allina Health COVID Research Registry or are receiving/have received therapy services for COVID-19 related sequelae at CKRI;
* English speaking
* Graduated from high school
* Able to see, hear, speak (with or without assistive devices)
* Access to computer or tablet and adequate internet connection to participate in video conference
* Has an email address;
* Own a smartphone with one of the following operating system versions:

iOS 9.0 - 9.3, 10.0 - 10.3, 12, 13.3, 13.7, 14.0 - 14.4 or later Android 8.0 - 8.1.0, 9, 10, 11 or later

* Agree to use personal smartphone to download mEMA application and respond to application notifications (mEMA is described in Sections 3.2.3.1 and 3.2.4.2.2);
* Willing and able to commit to attend all intervention sessions

Exclusion Criteria:

* History of neurologic disorder (such as stroke or brain injury) with residual impairments that likely interfere with learning;
* Any medical condition (physical or mental health) that interferes with the performance of everyday activities and roles.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2022-03-07 (Actual); Primary Completion 2023-03-07 (Actual); Study Completion 2024-01-22 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Wellbeing | Will be assessed at baseline (week 0) and completion (following session 8, week 12)
  Using the Psychological Scales of Wellbeing questionnaire (Ryff, 1989; Ryff, & Keyes, 1995), psychological wellbeing pre- and post- intervention will be tracked.

SECONDARY OUTCOMES:
Change in Meaning in Life Questionnaire | Will be assessed at baseline (week 0) and completion (following session 8, week 12)
  Meaning in Life Questionnaire (Steger et al., 2006): A 10-item questionnaire designed to measure 2 dimensions of meaning in life: Presence of Meaning (how much respondents feel their lives have meaning) and Search for Meaning (how much respondents strive to find meaning and understanding in their lives).
Change in Purpose Status Question | Will be assessed at baseline (week 0) and completion (following session 8, week 12)
  Purpose Status Question (PSQ) is a one-item questionnaire designed by the study team to measure participants' current purpose status

CONTACTS AND LOCATIONS:
Overall Officials: Mary V Radomski, OTR/L, PhD, Principal Investigator — Allina Health
Locations (1):
- Abbott Northwestern Hospital, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No
No IPD will be made available.